CLINICAL TRIAL: NCT02407990
Title: A Phase 1A/1B, Open Label, Multiple Dose, Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics and Antitumor Activities of the Anti-PD-1 Monoclonal Antibody BGB-A317 in Subjects With Advanced Tumors
Brief Title: Study of the Safety, Pharmacokinetics and Antitumor Activities of BGB-A317 in Participants With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317_Study_001
Record Dates: First submitted 2015-03-26; First posted 2015-04-03 (Estimated); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BGB-A317 Phase 1A (Experimental)
  Interventions: Biological: BGB-A317
- BGB-A317 Phase 1B (Experimental)
  Interventions: Biological: BGB-A317

INTERVENTIONS:
Biological: BGB-A317 — In the dose escalation part, the dose levels were escalated following a modified 3+3 dose escalation scheme. In the scheduled exploration part, participants were assigned to doses and dose schedules. In the fixed dose exploration part, participants were assigned to dose group(s) not to exceed the maximum tolerated dose. In the dose expansion part, participants were assigned to different groups based on their tumor type.
  Arms: BGB-A317 Phase 1A
Biological: BGB-A317 — Participants were assigned to different groups based on their tumor types
  Arms: BGB-A317 Phase 1B

SUMMARY:
This study evaluated the safety, tolerability, pharmacokinetic profile and treatment effect of a new drug known as BGB-A317 in participants with advanced tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must have had a histologically or cytologically confirmed advanced or metastatic tumor for which no effective standard therapy was available.

   1. For Phase 1A: no specific restriction
   2. For Phase 1B: histology specified below:

   i. non-small cell lung cancer (participants with documented epidermal growth factor receptor mutation or anaplastic lymphoma kinase rearrangement should have been excluded) ii. ovarian cancer iii. gastric cancer iv. hepatocellular carcinoma (HCC, Barcelona-Clinic Liver Cancer stage C, stage B not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach, and Child-Pugh A) v. head and neck squamous cell carcinoma vi. esophageal carcinoma vii. triple negative breast cancer viii. cholangiocarcinoma ix. renal cell cancer, bladder cancer, melanoma, Merkel-cell carcinoma, sarcoma, gastrointestinal stromal tumor, or cutaneous squamous cell carcinoma. Or any other solid tumors with known microsatellite instability-high or mismatch repair deficient status, such as colorectal cancer or pancreatic cancer
2. Participants with previously treated brain metastasis (es) that were asymptomatic or radiographically/clinically stable and not requiring steroids medications for 4 weeks prior to enrollment were permitted.
3. Participants must have had archival tumor tissues or agreed to a tumor biopsy for analysis of predictive biomarkers such as programmed death-ligand 1 (PD-L1). (Fresh tumor biopsies were strongly recommended at baseline for biomarker analysis in participants with readily accessible tumor lesions and who consented to the biopsies).
4. Participants must have had measurable disease as defined per Response Evaluation Criteria in Solid Tumor Version 1.1.
5. Eastern Cooperative Oncology Group performance status of ≤ 1.
6. Participants must have had adequate organ function as indicated by the following laboratory values:

   * Absolute neutrophil count ≥ 1,500 /microliter
   * Platelets ≥ 100,000 / milliliter (mL)
   * Hemoglobin ≥ 9 grams/deciliter or ≥ 5.6 millimoles/liter
   * Serum creatinine ≤ 1.5 X upper limit of normal (ULN)
   * Serum total bilirubin ≤ 1.5 X ULN
   * Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) and alanine aminotransferase (serum glutamic pyruvic transaminase) ≤ 2.5 X ULN or ≤ 5 X ULN for participants with liver metastases
   * International normalized ratio or prothrombin time ≤ 1.5 X ULN
   * Activated partial thromboplastin time ≤ 1.5 X ULN

Key Exclusion Criteria:

1. History of severe hypersensitivity reactions to other Monoclonal antibodies.
2. Prior malignancy active within the previous 2 years except for tumor for which a participant was enrolled in the study, and locally curable cancers that had been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
3. Prior therapies targeting PD-1 or PD-L1.
4. Participants who failed to meet enrollment criteria for other PD-1 or PD-L1 trials solely due to low or negative predictive biomarkers.
5. Participants with active autoimmune diseases or history of autoimmune diseases should have been excluded.
6. Participants should have been excluded if they had a condition requiring systemic treatment with either corticosteroids (> 10 milligrams daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
7. Had history of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies.
8. Known history of human immunodeficiency virus.
9. Active infection requiring therapy, positive tests for hepatitis B surface antigen or hepatitis C ribonucleic acid except in participant with HCC, who met the following criteria:

   * Hepatitis B virus (HBV) viral load < 200 international units/mL (approximately 1000 combined positive score/mL)
   * Participants with active HBV infection needed to be on anti-HBV suppression ≥ 3 months, throughout treatment and for 6 months after
   * Participants hepatitis C virus (HCV)-positive after successful treatment (defined as sustained virologic response [SVR] 12 or SVR 24) were allowed as long as 4 weeks had passed between completion of HCV therapy and start of study drug
10. Use of any vaccines against infectious diseases (for example, influenza, varicella) within 4 weeks (28 days) of initiation of study therapy and 60 days after the last administration of the study medication.

Note: Other protocol defined Inclusion/Exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (27):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Oncology Consultants, P.A., Houston, Texas
- Australia (13):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Tasman Oncology Research Ltd, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Health Hospital, Heidelberg, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Linear Clinical Research/Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (3):
  - Auckland City Hospital, Grafton
  - Waikato, Hamilton
  - Wellington Hospital, Wellington
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
  - Chang Gung Memorial Hospital, Sachin, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Desai J, Deva S, Lee JS, Lin CC, Yen CJ, Chao Y, Keam B, Jameson M, Hou MM, Kang YK, Markman B, Lu CH, Rau KM, Lee KH, Horvath L, Friedlander M, Hill A, Sandhu S, Barlow P, Wu CY, Zhang Y, Liang L, Wu J, Paton V, Millward M. Phase IA/IB study of single-agent tislelizumab, an investigational anti-PD-1 antibody, in solid tumors. J Immunother Cancer. 2020 Jun;8(1):e000453. doi: 10.1136/jitc-2019-000453. PMID 32540858
- [Derived] Ye D, Desai J, Shi J, Liu SM, Shen W, Liu T, Shi Y, Wang D, Liang L, Yang S, Ma X, Jin W, Zhang P, Huang R, Shen Z, Zhang Y, Wu YL. Co-enrichment of CD8-positive T cells and macrophages is associated with clinical benefit of tislelizumab in solid tumors. Biomark Res. 2023 Mar 7;11(1):25. doi: 10.1186/s40364-023-00465-w. PMID 36879284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 27 centers in 5 countries, enrolled from June 2015 to October 2017 across both Phases, and was initiated in June 2015. After a 5-year period the sponsor decided to close the study as primary and secondary endpoints were met. Participants still on treatment were rolled into a separate long-term extension study (BGB-A317-290-LTE1) to continue treatment.
Groups:
- BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg: Participants were dosed at 0.5 milligrams/kilograms (mg/kg), tislelizumab, once every 2 weeks (Q2W) until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration.
- BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg: Participants were dosed at 2.0 mg/kg tislelizumab, Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration.
- BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg: Participants were dosed at 5.0 mg/kg tislelizumab, Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration.
- BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg: Participants were dosed at 10.0 mg/kg tislelizumab, Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration.
- BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg: Participants received selected dosing based on Part 1 of 2.0 mg/kg tislelizumab, once every 3 weeks (Q3W) until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
- BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg: Participants received selected dosing based on Part 1 of 5.0 mg/kg tislelizumab,Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
- BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg: Participants received selected maximum tolerated dose of 200.0 mg/kg tislelizumab, Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
- BGB-A317 Phase 1B: Participants were dosed at 5 mg/kg tislelizumab, Q3W until confirmed disease progression, intolerable toxicity, subject discontinuation/ withdrawal or at the discretion of the Investigator in consultation with Sponsor, as determined by the safety monitoring committee, in 9 indication expansion Arms. Each treatment cycle was 21 days in duration.
Period: Overall Study
Arm/Group | BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg | BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg | BGB-A317 Phase 1B
Started | 3 | 26 | 26 | 7 | 21 | 20 | 13 | 335
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 26 | 26 | 7 | 21 | 20 | 13 | 335
Not completed — Death | 2 | 22 | 23 | 7 | 17 | 16 | 10 | 248
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 17
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 30
Not completed — Study Terminated by Sponsor | 1 | 3 | 3 | 0 | 3 | 4 | 3 | 37
Not completed — Logistics | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Rolled into long-term extension study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg: Participants were dosed at 0.5 milligrams/kilograms (mg/kg), once every 2 weeks (Q2W) until death, disease progression, unacceptable toxicities, or withdrawal of consent.. Each treatment cycle was 28 days in duration.
- BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg: Participants were dosed at 2.0 mg/kg, Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration
- BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg: Participants were dosed at 5.0 mg/kg, Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent.. Each treatment cycle was 28 days in duration
- BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg: Participants were dosed at 10.0 mg/kg, Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration.
- BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg: Participants received selected dosing based on Part 1 of 2.0 mg/kg once every 3 weeks (Q3W) until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
- BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg: Participants received selected dosing based on Part 1 of 5.0 mg/kg Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
- BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg: Participants received selected maximum tolerated dose of 200.0 mg/kg Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
- BGB-A317 Phase 1B: Participants were dosed at 5 mg/kg Q3W until confirmed disease progression, intolerable toxicity, subject discontinuation/ withdrawal or at the discretion of the Investigator in consultation with Sponsor, as determined by the safety monitoring committee, in 9 indication expansion Arms. Each treatment cycle was 21 days in duration.
- Total: Total of all reporting groups
Arm/Group | BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg | BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg | BGB-A317 Phase 1B | Total
Number analyzed (Participants) | 3 | 26 | 26 | 7 | 21 | 20 | 13 | 335 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (7.02) | 59.1 (11.15) | 57.8 (13.32) | 57.1 (8.13) | 63.6 (10.09) | 62.6 (11.14) | 58.4 (17.76) | 59.5 (11.92) | 59.6 (11.96)
Age, Customized [Count of Participants; unit: Participants]
  < 65 Years | 3 | 18 | 16 | 6 | 8 | 11 | 6 | 217 | 285
  ≥ 65 Years | 0 | 8 | 10 | 1 | 13 | 9 | 7 | 118 | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15 | 4 | 10 | 12 | 5 | 144 | 205
  Male | 0 | 14 | 11 | 3 | 11 | 8 | 8 | 191 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 8 | 10
  Not Hispanic or Latino | 3 | 24 | 26 | 7 | 21 | 20 | 13 | 322 | 436
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 2 | 3 | 0 | 1 | 3 | 1 | 120 | 130
  Chinese (enrolled from Taiwan sites) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 61
  Non-Chinese | 0 | 2 | 3 | 0 | 1 | 3 | 1 | 59 | 69
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  White | 3 | 22 | 23 | 7 | 19 | 16 | 11 | 189 | 290
  Other | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 18 | 23

OUTCOME MEASURES:

1. Primary Outcome: Phase 1A: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of an investigational product. All AEs were monitored per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version [v] 4.03 2010).
Time Frame: Day -28 through 5 years and 2 months
Population: Safety Analysis Set (SAF) included all participants who had received any dose of tislelizumab. The analysis was pre-specified to be a pooled analysis of all Part 1A cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- BGB-A317 Phase 1A: In Part 1, participants were dosed at 0.5 mg/kg, 2 mg/kg, 5 mg/kg, and 10 mg/kg Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration. In Part 2, participants received selected dosing based on Part 1 at Q2W and/or Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days and 21 days in duration, respectively. In Part 3: participants received a fixed dose that did not exceed the selected maximum tolerated dose (MTD), which was 200 mg Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants | 114

2. Primary Outcome: Phase 1A: Number Of Participants With Abnormal Physical Examination Values
Description: A complete physical examination, vital signs (systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse rate, temperature, and respiratory rate), and weight were performed pre-specified time points for Phase 1A. During the treatment period, symptom-directed physical examinations were performed. If there were no complaints and no abnormal findings from the previous visit for a particular organ system, a physical examination of that organ system was not required.
Time Frame: Day 1 and Day 15 of each cycle through 30 (+/- 7) days after last dose (up to 5 years and 2 months)
Population: Safety Analysis Set: all participants who had received any dose of tislelizumab. The analysis was pre-specified to be a pooled analysis of all Part 1A cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- BGB-A317 Phase 1A: In Part 1, participants were dosed at 0.5 mg/kg, 2 mg/kg, 5 mg/kg, and 10 mg/kg Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration. In Part 2, participants received selected dosing based on Part 1 at Q2W and/or Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days and 21 days in duration, respectively. In Part 3: participants received a fixed dose that did not exceed the selected MTD, which was 200 mg Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants
  At least one postbaseline pulse rate measure ≤ 45 beats per minute (bpm) | 1
  At least one postbaseline pulse rate measure ≥ 120 bpm | 6
  At least one postbaseline SBP measure ≤ 60 millimeters of mercury (mmHg) | 0
  At least one postbaseline SBP measure ≤ 90 mmHg | 9
  At least one postbaseline SBP measure ≥ 160 mmHg | 17
  At least one postbaseline DBP measure ≥ 100 mmHg | 5

3. Primary Outcome: Phase 1A: Number Of Participants Experiencing Dose-dependent Toxicity Through Ophthalmology Findings
Description: Ophthalmological examinations (such as eyesight/visual acuity, fundoscopy, slit lamp microscopy, and optical coherence tomography [or equivalent diagnostic test]) were performed at pre-specified time points for Phase 1A. Eye exam, visual acuity test, and optical coherence tomography (or equivalent diagnostic test) will be assessed by an appropriate specialist at Screening. Participants dosed underwent subsequent ophthalmologic examinations, a specified in the protocol, by an appropriate specialist during study treatment.
Time Frame: Day 15 of cycle 1, Day 1 of Cycle 2 and all additional cycles, and 30 (+/- 7) days after last dose (up to 5 years and 2 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants | 0

4. Primary Outcome: Phase 1A: Number Of Participants With Abnormal Electrocardiograms
Description: Electrocardiograms were obtained at pre-specified time points. Significant QT interval corrected for heart rate (QTc) prolongation was defined as an interval ≥ 500 milliseconds (msec) or an interval which increases by ≥ 60 msec over baseline.
Time Frame: Days 1 and 15 of cycle 1; Day 1 of cycle 2 and all additional cycles; Day 1 of cycle 4; 30 (+/- 7) days after last dose (up to 5 years and 2 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants
  At least 1 postbaseline QT corrected using Fridericia's formula (QTcF) Interval measure of >450 msec | 31
  At least 1 postbaseline QTcF Interval measure of > 480 msec | 9
  At least 1 postbaseline QTcF Interval measure of > 500 msec | 3
  At least 1 postbaseline QTcF Interval measure ≤ 30 msec increase from baseline | 73
  At least 1 postbaseline QTcF Interval measure ≤ 30 and ≤ 60 msec increase from baseline | 35
  At least 1 postbaseline QTcF Interval measure > 60 msec increase from baseline | 8

5. Primary Outcome: Phase 1A: Number Of Participants With Abnormal Laboratory Values
Description: Clinical chemistry, hematology, coagulation, and urinalysis were performed at pre-specified time points for Phase 1A. If warranted, additional testing was done, or the relevant tests done more frequently in accordance with institutional guidelines. All participants who had any Grade 3 or Grade 4 laboratory abnormalities at withdrawal from the study were followed up until they had returned to Grade 1 or Grade 2, unless these were not likely to improve due to the underlying disease. Participants experiencing decreases (low) and increases (high) to ≥ Grade 3 are reported.
Time Frame: Day -28 (predose), Days 1, 8, and 15 of cycle 1; Days 1 and 15 of cycle 2 and additional cycles; Days 1 and 15 of cycle 4; 30 (+/- 7) days after last dose (up to 5 years and 2 months)
Population: Safety Analysis Set: participants who had received any dose of tislelizumab and with baseline assessment and at least one post-baseline assessment. The analysis was pre-specified to be a pooled analysis of all Part 1A cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants
  Alanine Aminotransferase: High | 6
  Albumin: Low | 11
  Alkaline Phosphatase: High | 7
  Aspartate Aminotransferase: High | 5
  Bilirubin: High | 7
  Calcium: Low | 7
  Calcium: High | 2
  Creatinine: High | 6
  Glucose: Low | 5
  Glucose: High | 13
  Hemoglobin: Low | 6
  Leukocytes: Low | 3
  Leukocytes: High | 0
  Lymphocytes: Low | 22
  Lymphocytes: High | 2
  Neutrophils: Low | 2
  Phosphate: Low | 19
  Platelets: Low | 1
  Potassium: Low | 21
  Potassium: High | 7
  Sodium: Low | 8
  Sodium: High | 0

6. Primary Outcome: Phase 1A: Number Of Participants Experiencing Severe AEs
Description: All AEs were monitored per the NCI-CTCAE (v 4.03 2010). In addition to performing the CTCAE assessment, the intensity of each AE and serious adverse event (SAE) recorded was assigned to one of the following categories based on the Investigator's clinical judgment: Mild: an event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; moderate: An event that is sufficiently discomforting to interfere with normal everyday activities; severe: An event that prevents normal everyday activities. Severity was a category utilized for rating the intensity of an event and, accordingly, both AEs and SAEs could be assessed as severe.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants | 14

7. Primary Outcome: Phase 1B: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants in the study whose best overall response was either complete response (CR) or partial response (PR) as assessed by investigators based on Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1.
Time Frame: Day -28 through 5 years and 2 months
Population: Efficacy Evaluable Set (EFF) included all participants in the SAF with measurable disease at baseline per RECIST v 1.1 who had at least 1 evaluable post-baseline tumor assessment, unless discontinued due to clinical disease progression, or death within 10 weeks of the first dose date.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BGB-A317 Phase 1B: Participants were dosed at 5 mg/kg Q3W until confirmed disease progression, intolerable toxicity, participant discontinuation/ withdrawal or at the discretion of the Investigator in consultation with Sponsor, as determined by the safety monitoring committee, in 9 indication expansion Arms. Each treatment cycle was 21 days in duration.
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
percentage of participants | 11.6 [8.41 to 15.57]

8. Secondary Outcome: Phase 1A: Area Under The Plasma Concentration-time Curve Within the Dosing Interval (AUC0-tau) For Tislelizumab
Time Frame: Cycle 1 Day 1-1 hour pre-dose, End of infusion, 1, 5, 6, 24, and 72 hours post-dose; Day 15 and Cycle 2 Day 1 Pre-dose
Population: PK Analysis Set (PKS) included participants who had received at least the first dose of tislelizumab and provided PK samples as per protocol following first dosing.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter*day
Arm/Group | BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg | BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 18 | 20 | 12
micrograms/milliliter*day | 84.92 (35.90) | 332.2 (57.33) | 811.8 (239.5) | 1916.0 (458.5) | 512.1 (122.2) | 1219.0 (287.4) | 674.7 (173.6)

9. Secondary Outcome: Phase 1A: Maximum Observed Plasma Concentration (Cmax) For Tislelizumab
Time Frame: Cycle 1 Day 1-1 hour pre-dose, End of infusion, 1, 5, 6, 24, and 72 hours post-dose; Day 15 and Cycle 2 Day 1 Pre-dose
Population: PKS included participants who had received at least the first dose of tislelizumab and provided PK samples as per protocol following first dosing.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg | BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 18 | 20 | 12
micrograms/milliliter | 13.5 (3.80) | 48.3 (6.89) | 147.0 (50.8) | 278.0 (53.7) | 56.8 (12.8) | 130.0 (29.7) | 77.2 (13.9)

10. Secondary Outcome: Phase 1A: Time To Maximum Concentration (Tmax) For Tislelizumab
Time Frame: Cycle 1 Day 1-1 hour pre-dose, End of infusion, 1, 5, 6, 24, and 72 hours post-dose; Day 15 and Cycle 2 Day 1 Pre-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Groups:
- BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg: Participants were dosed at 0.5 milligrams/kilograms (mg/kg), tislelizumab, once every 2 weeks (Q2W). until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration.
Arm/Group | BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg | BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 18 | 20 | 12
hours | 3.46 (3.12) | 2.39 (0.89) | 2.48 (0.73) | 2.43 (1.83) | 1.57 (0.65) | 4.95 (15.4) | 1.40 (0.82)

11. Secondary Outcome: Phase 1A: Half-life (T½) For Tislelizumab
Time Frame: Cycle 1 Day 1-1 hour pre-dose, End of infusion, 1, 5, 6, 24, and 72 hours post-dose; Day 15 and Cycle 2 Day 1 Pre-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Groups:
- BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg: Participants received selected dosing based on Part 1 of 2.0 mg/kg tislelizumab, once every 3 weeks (Q3W). until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 21 days in duration.
Arm/Group | BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg | BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 18 | 20 | 12
hours | 10.7 (3.90) | 12.9 (1.2) | 15.0 (14.4) | 14.5 (4.04) | 17.1 (8.14) | 19.6 (7.63) | 16.8 (5.50)

12. Secondary Outcome: Phase 1A - Part 3: Clearance (Cl) For Tislelizumab
Time Frame: Cycle 1 Day 1-1 hour pre-dose, End of infusion, 1, 5, 6, 24, and 72 hours post-dose; Day 15 and Cycle 2 Day 1 Pre-dose
Population: PK Analysis Set (PKS) included participants who had received at least the first dose of tislelizumab and provided PK samples as per protocol following first dosing. per-pre-specification, data was analyzed only for Part 3 of Phase 1A.
Measure: Geometric Mean (95% Confidence Interval); unit: liters/day
Arm/Group | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg
Number analyzed (Participants) | 12
liters/day | 0.186 [0.135 to 0.256]

13. Secondary Outcome: Phase 1A/1B: Number Of Participants With Anti-drug Antibodies (ADAs)
Description: Immunogenicity was summarized by the number and percentage of participants who developed detectable treatment-emergent ADAs, which included positive ADAs and neutralizing antibodies (NAb).
Time Frame: Day 1 of Cycles 1 through 15
Population: Evaluable set: participants who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result.
Measure: Number; unit: Participants
Groups:
- BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg: Participants were dosed at 0.5 milligrams/kilograms (mg/kg), once every 2 weeks (Q2W) until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration.
- BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg: Participants were dosed at 5.0 mg/kg, Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration
- BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg and BGB-A317 Phase 1B: Phase 1A: Participants received selected dosing based on Part 1 of 5.0 mg/kg Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent.. Each treatment cycle was 21 days in duration.
  Phase 1B; Participants were dosed at 5 mg/kg Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent, as determined by the safety monitoring committee, in 9 indication expansion Arms. Each treatment cycle was 21 days in duration.
Arm/Group | BGB-A317 Phase 1A - Part 1 - 0.5 mg/kg | BGB-A317 Phase 1A - Part 1 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 5.0 mg/kg | BGB-A317 Phase 1A - Part 1 - 10.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 2.0 mg/kg | BGB-A317 Phase 1A - Part 2 - 5.0 mg/kg and BGB-A317 Phase 1B | BGB-A317 Phase 1A - Part 3 - 200.0 mg/kg
Number analyzed (Participants) | 3 | 21 | 25 | 6 | 19 | 285 | 11
Participants | 1 | 6 | 5 | 1 | 6 | 43 | 3

14. Secondary Outcome: Phase 1A: ORR
Description: The ORR was defined as the percentage of participants in the study whose best overall response was either CR or PR as assessed by investigators based on RECIST v 1.1.
Time Frame: Day -28 through 5 years and 2 months
Population: Efficacy Evaluable Set included all participants in the SAF with measurable disease at baseline per RECIST v 1.1 who had at least 1 evaluable post-baseline tumor assessment, unless discontinued due to clinical disease progression, or death within 10 weeks of the first dose date. The analysis was pre-specified to be a pooled analysis of all Part 1A cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
percentage of participants | 18.1 [11.57 to 26.33]

15. Secondary Outcome: Phase 1A: CR Rate
Description: The CR rate was based on RECIST v 1.1 and the results of Investigator evaluations.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants | 6

16. Secondary Outcome: Phase 1A: PR Rate
Description: The PR rate was based on RECIST v 1.1 and the results of Investigator evaluations.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants | 15

17. Secondary Outcome: Phase 1A: Stable Disease (SD) Rate
Description: The SD rate was based on RECIST v 1.1 and the results of Investigator evaluations.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
Participants | 42

18. Secondary Outcome: Phase 1A: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of first study dose to disease progression or death whichever occurs first. Participants without an event (no disease progression or death) were censored at the date of "last tumor assessment". Participants with no baseline or post-baseline tumor assessments were censored at Day 1. PFS was based on RECIST v 1.1 and the results of Investigator evaluations.
Time Frame: Day -28 through 5 years and 2 months
Population: Efficacy Evaluable Set included all participants in the SAF with measurable disease at baseline per RECIST v 1.1 who had at least 1 evaluable post-baseline tumor assessment, unless discontinued due to clinical disease progression, or death within 10 weeks of the first dose date.The analysis was pre-specified to be a pooled analysis of all Part 1A cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
months | 3.5 [2.1 to 3.8]

19. Secondary Outcome: Phase 1A: Overall Survival (OS)
Description: OS was defined as the time interval between the date of the first study drug dose to the date of death for any cause. Kaplan-Meier methodology was used to estimate OS at various time points. The OS was based on RECIST v 1.1 and the results of Investigator evaluations.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
months | 13.6 [9.9 to 17.5]

20. Secondary Outcome: Phase 1A: Duration Of Response (DOR)
Description: DOR for responders (CR or PR) was defined as the time interval between the date of the earliest qualifying response and the date of progressive disease or death for any cause, whichever occurred earlier. For participants who were alive without progression following the qualifying response, DOR was censored on the date of last evaluable tumor assessment or last follow-up for progression of disease. The DOR was based on RECIST v 1.1 and the results of Investigator evaluations.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGB-A317 Phase 1A
Number analyzed (Participants) | 116
months | 14.6 [8.3 to NA] — NA = Not estimable due to insufficient number of participants with events

21. Secondary Outcome: Phase 1B: Number of Participants Experiencing AEs
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of an investigational product. All AEs were monitored per the NCI-CTCAE (v 4.03 2010).
Time Frame: Day -28 through 5 years and 2 months
Population: Safety Analysis Set (SAF) included all patients who had received any dose of tislelizumab
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
Participants | 322

22. Secondary Outcome: Phase 1B: Steady State Plasma Trough Concentration Of Tislelizumab
Time Frame: Pre-dose, Day 1 Cycle 5 and every other Cycle in the first 6 months, every 4 cycles in the next 6 months, once every 6 months up to end of treatment (up to 5 years and 2 months)
Population: PK Analysis Set included participants who had received at least the first dose of tislelizumab and provided PK samples as per protocol following first dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 145
micrograms/milliliter
  Non-Small Cell Lung Cancer: number analyzed (Participants) | 30
  Non-Small Cell Lung Cancer | 63.9 (47.8)
  Ovarian Cancer: number analyzed (Participants) | 10
  Ovarian Cancer | 90.4 (66.7)
  Gastric Cancer: number analyzed (Participants) | 15
  Gastric Cancer | 40.7 (91.4)
  Hepatocellular Carcinoma: number analyzed (Participants) | 27
  Hepatocellular Carcinoma | 54.4 (56.8)
  Head & Neck Squamous Cell Carcinoma: number analyzed (Participants) | 11
  Head & Neck Squamous Cell Carcinoma | 77.4 (45.8)
  Esophageal Carcinoma: number analyzed (Participants) | 18
  Esophageal Carcinoma | 57.8 (62.4)
  Triple Negative Breast Cancer: number analyzed (Participants) | 3
  Triple Negative Breast Cancer | 47.8 (78.9)
  Cholangio Carcinoma: number analyzed (Participants) | 7
  Cholangio Carcinoma | 65.7 (47.9)
  Other Solid Tumors: number analyzed (Participants) | 24
  Other Solid Tumors | 80.4 (43.5)

23. Secondary Outcome: Phase 1B: PFS
Description: as for outcome 18
Time Frame: Day -28 through 5 years and 2 months
Population: Efficacy Evaluable Set included all participants in the SAF with measurable disease at baseline per RECIST v 1.1 who had at least 1 evaluable post-baseline tumor assessment, unless discontinued due to clinical disease progression, or death within 10 weeks of the first dose date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
months | 2.1 [2.0 to 2.2]

24. Secondary Outcome: Phase 1B: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of participants who achieve CR, PR, and SD based on RECIST v 1.1 in participants with select tumor types.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
percentage of participants | 41.2 [35.87 to 46.67]

25. Secondary Outcome: Phase 1B: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of participants who achieved CR, PR, and durable SD [SD ≥24 weeks] based on RECIST v 1.1 in participants with select tumor types.
Time Frame: Day -28 through 5 years and 2 months
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
percentage of participants | 24.5 [19.97 to 29.45]

26. Secondary Outcome: Phase 1B: Number Of Participants With Abnormal Physical Examination Values
Description: A complete physical examination, vital signs (SBP, DBP, pulse rate, temperature, and respiratory rate), and weight were performed pre-specified time points for Phase 1B. During the treatment period, symptom-directed physical examinations were performed. If there were no complaints and no abnormal findings from the previous visit for a particular organ system, a physical examination of that organ system was not required.
Time Frame: Day -28 (predose), Days 1, 4, 8, and 15 of cycle 1; Day 1 of cycle 2; through 30 (+/- 7) days after last dose up to 5 years and 2 months
Population: Safety Analysis Set: all participants who had received any dose of tislelizumab and with baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
Participants
  At least one postbaseline pulse rate measure ≤ 45 bpm: number analyzed (Participants) | 312
  At least one postbaseline pulse rate measure ≤ 45 bpm | 5
  At least one postbaseline pulse rate measure ≥ 120 bpm: number analyzed (Participants) | 312
  At least one postbaseline pulse rate measure ≥ 120 bpm | 26
  At least one postbaseline SBP measure ≤ 60 mmHg: number analyzed (Participants) | 312
  At least one postbaseline SBP measure ≤ 60 mmHg | 1
  At least one postbaseline SBP measure ≤ 90 mmHg: number analyzed (Participants) | 312
  At least one postbaseline SBP measure ≤ 90 mmHg | 24
  At least one postbaseline SBP measure ≥ 160 mmHg: number analyzed (Participants) | 312
  At least one postbaseline SBP measure ≥ 160 mmHg | 30
  At least one postbaseline DBP measure ≥ 100 mmHg: number analyzed (Participants) | 312
  At least one postbaseline DBP measure ≥ 100 mmHg | 12

27. Secondary Outcome: Phase 1B: Number Of Participants Experiencing Dose-dependent Toxicity Through Ophthalmology Findings
Description: Ophthalmological examinations (such as eyesight/visual acuity, fundoscopy, slit lamp microscopy, and optical coherence tomography [or equivalent diagnostic test]) were performed at pre-specified time points for Phase 1B. Eye exam, visual acuity test, and optical coherence tomography (or equivalent diagnostic test) will be assessed by an appropriate specialist at Screening. Participants dosed underwent subsequent ophthalmologic examinations, a specified in the protocol, by an appropriate specialist during study treatment.
Time Frame: Day -28 (predose), Day 1 of cycle 2 and additional cycles, and 30 (+/- 7) days after last dose up to 5 years and 2 months
Population: Safety Analysis Set (SAF) included all patients who had received any dose of tislelizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
Participants | 0

28. Secondary Outcome: Phase 1B: Number Of Participants With Abnormal Electrocardiograms
Description: Electrocardiograms were obtained at pre-specified time points. Significant QTc prolongation was defined as an interval ≥ 500 msec or an interval which increases by ≥ 60 msec over baseline.
Time Frame: Day -28 (predose), Days 1 and 15 of cycle 1; Day 1 of cycle 2 and additional cycles; 30 (+/- 7) days after last dose up to 5 years and 2 months
Population: Safety Analysis Set: all participants who had received any dose of tislelizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
Participants
  At least 1 postbaseline QTcF Interval measure > 450 msec: number analyzed (Participants) | 312
  At least 1 postbaseline QTcF Interval measure > 450 msec | 84
  At least 1 postbaseline QTcF Interval measure > 480 msec: number analyzed (Participants) | 312
  At least 1 postbaseline QTcF Interval measure > 480 msec | 24
  At least 1 postbaseline QTcF Interval measure > 500 msec: number analyzed (Participants) | 312
  At least 1 postbaseline QTcF Interval measure > 500 msec | 10
  At least 1 postbaseline QTcF Interval measure ≤ 30 msec increase from baseline: number analyzed (Participants) | 312
  At least 1 postbaseline QTcF Interval measure ≤ 30 msec increase from baseline | 241
  At least 1 postbaseline QTcF Interval measure >30 and ≤ 60 msec increase from baseline: number analyzed (Participants) | 312
  At least 1 postbaseline QTcF Interval measure >30 and ≤ 60 msec increase from baseline | 67
  At least 1 postbaseline QTcF Interval measure > 60 msec increase: number analyzed (Participants) | 312
  At least 1 postbaseline QTcF Interval measure > 60 msec increase | 22

29. Secondary Outcome: Phase 1B: Number Of Participants With Abnormal Laboratory Values
Description: Clinical chemistry, hematology, coagulation, and urinalysis will be performed at pre-specified time points for Phase 1A and Phase 1B respectively. If warranted, additional testing was done, or the relevant tests done more frequently in accordance with institutional guidelines. All participants who had any Grade 3 or Grade 4 laboratory abnormalities at withdrawal from the study were followed up until they had returned to Grade 1 or Grade 2, unless these were not likely to improve due to the underlying disease. Participants experiencing decreases (low) and increases (high) to ≥ Grade 3 are reported.
Time Frame: Day -28 (predose), Days 1, 8, and 15 of cycle 1; Day 1 of cycle 2 and additional cycles; 30 (+/- 7) days after last dose up to 5 years and 2 months
Population: Safety Analysis Set: participants who had received any dose of tislelizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
Participants
  Alanine Aminotransferase: High | 21
  Albumin: Low | 42
  Alkaline Phosphatase: High | 21
  Aspartate Aminotransferase: High | 21
  Bilirubin: High | 22
  Calcium: Low | 12
  Calcium: High | 7
  Creatinine: High | 20
  Glucose: Low | 8
  Glucose: High | 32
  Hemoglobin: Low | 19
  Leukocytes: Low | 8
  Leukocytes: High | 1
  Lymphocytes: Low: number analyzed (Participants) | 223
  Lymphocytes: Low | 33
  Lymphocytes: High: number analyzed (Participants) | 223
  Lymphocytes: High | 2
  Neutrophils: Low: number analyzed (Participants) | 223
  Neutrophils: Low | 5
  Phosphate: Low | 42
  Platelets: Low | 3
  Potassium: Low | 35
  Potassium: High | 4
  Sodium: Low | 25
  Sodium: High | 1

30. Secondary Outcome: Phase 1B: Number Of Participants Experiencing Severe AEs
Description: All AEs were monitored per the NCI-CTCAE (v 4.03 2010). In addition to performing the CTCAE assessment, the intensity of each AE and SAE recorded was assigned to one of the following categories based on the Investigator's clinical judgment: Mild: an event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; moderate: An event that is sufficiently discomforting to interfere with normal everyday activities; severe: An event that prevents normal everyday activities. Severity was a category utilized for rating the intensity of an event and, accordingly, both AEs and SAEs could be assessed as severe.
Time Frame: Day -28 through 5 years and 2 months
Population: Safety Analysis Set (SAF) included all patients who had received any dose of tislelizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-A317 Phase 1B
Number analyzed (Participants) | 335
Participants | 27

ADVERSE EVENTS:
Time Frame: Day -28 through 5 years and 2 months
Description: The analysis was pre-specified to be a pooled analysis of all Part 1A cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Groups:
- BGB-A317 Phase 1A: In Part 1, participants were dosed at 0.5 mg/kg, 2 mg/kg, 5 mg/kg, and 10 mg/kg Q2W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days in duration. In Part 2, participants received selected dosing based on Part 1 at Q2W and/or Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent. Each treatment cycle was 28 days and 21 days in duration, respectively. In Part 3: participants received a fixed dose that did not exceed the selected MTD, which is 200 mg Q3W until death, disease progression, unacceptable toxicities, or withdrawal of consent.. Each treatment cycle was 21 days in duration.
Arm/Group | BGB-A317 Phase 1A | BGB-A317 Phase 1B
All-Cause Mortality (participants affected / at risk) | 97/116 | 249/335
Serious Adverse Events (participants affected / at risk) | 40/116 | 131/335
Other Adverse Events (participants affected / at risk) | 112/116 | 302/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BGB-A317 Phase 1A (N=116) | BGB-A317 Phase 1B (N=335)
Vomiting (Gastrointestinal disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Ascites (Gastrointestinal disorders) | 2 | 4
Colitis (Gastrointestinal disorders) | 3 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 2 | 3
Pyrexia (General disorders) | 2 | 6
Pneumonia (Infections and infestations) | 4 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 2
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastric varices (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 3
Cholangitis (Hepatobiliary disorders) | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 0 | 4
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 0 | 2
Acute sinusitis (Infections and infestations) | 1 | 0
Bacterascites (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Bone tuberculosis (Infections and infestations) | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Complicated appendicitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Orbital infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Thoracic radiculopathy (Nervous system disorders) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BGB-A317 Phase 1A (N=116) | BGB-A317 Phase 1B (N=335)
Nausea (Gastrointestinal disorders) | 41 | 71
Diarrhoea (Gastrointestinal disorders) | 33 | 49
Constipation (Gastrointestinal disorders) | 28 | 51
Abdominal pain (Gastrointestinal disorders) | 25 | 42
Vomiting (Gastrointestinal disorders) | 19 | 42
Abdominal pain upper (Gastrointestinal disorders) | 9 | 19
Abdominal distension (Gastrointestinal disorders) | 6 | 17
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 17
Dry mouth (Gastrointestinal disorders) | 6 | 11
Dysphagia (Gastrointestinal disorders) | 3 | 11
Ascites (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Mouth ulceration (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 47 | 80
Pyrexia (General disorders) | 7 | 31
Oedema peripheral (General disorders) | 13 | 24
Non-cardiac chest pain (General disorders) | 9 | 12
Influenza like illness (General disorders) | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 40
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 23
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 21
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Rash (Skin and subcutaneous tissue disorders) | 23 | 39
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 38
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 12
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 20 | 74
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 17
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 35
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 12
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 15 | 28
Urinary tract infection (Infections and infestations) | 8 | 22
Oral candidiasis (Infections and infestations) | 8 | 17
Lower respiratory tract infection (Infections and infestations) | 4 | 11
Pneumonia (Infections and infestations) | 4 | 9
Nasopharyngitis (Infections and infestations) | 4 | 7
Oral herpes (Infections and infestations) | 4 | 2
Weight decreased (Investigations) | 5 | 35
Alanine aminotransferase increased (Investigations) | 9 | 17
Aspartate aminotransferase increased (Investigations) | 4 | 18
Blood creatinine increased (Investigations) | 7 | 12
Headache (Nervous system disorders) | 9 | 28
Dizziness (Nervous system disorders) | 10 | 12
Lethargy (Nervous system disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 5 | 29
Anxiety (Psychiatric disorders) | 8 | 6
Hypothyroidism (Endocrine disorders) | 8 | 22
Hyperthyroidism (Endocrine disorders) | 5 | 14
Anaemia (Blood and lymphatic system disorders) | 12 | 28
Infusion related reaction (Injury, poisoning and procedural complications) | 12 | 13
Hot flush (Vascular disorders) | 4 | 6
Hypotension (Vascular disorders) | 5 | 5
Proteinuria (Renal and urinary disorders) | 3 | 14
Dry eye (Eye disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT02407990/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT02407990/SAP_001.pdf